CLINICAL TRIAL: NCT02444598
Title: A Prospective, Randomized, Controlled Trial of Negative-pressure Wound Therapy Use in Conflict-related Extremity Wounds (VACoCREW Trial)
Brief Title: Trial of Negative-pressure Wound Therapy Use in Conflict-related Extremity Wounds
Acronym: VACoCREW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); Jordan University of Science and Technology (Other); Stockholm South General Hospital (Other); Center for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Jonas Malmstedt, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KISOS001
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Wounds, Gunshot; Arm Injuries; Leg Injuries; Wound Infection
Keywords: wounds; negative-pressure wound therapy; conflict; gunshot wound; blast injuries; civilian; war
MeSH Terms: conditions — Wounds, Gunshot; Arm Injuries; Leg Injuries; Wound Infection; Wounds and Injuries; Blast Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative-pressure wound therapy (Experimental): Vaccum Assisted Closure device. Patients will receive negative-pressure wound therapy according to manufacturer treatment guidelines.
  Interventions: Device: Vaccum Assisted Closure device
- Standard (Active Comparator): Patients will be treated with conventional wound dressings according to local treatment protocols.
  Interventions: Procedure: Conventional wound dressings

INTERVENTIONS:
Device: Vaccum Assisted Closure device — Negative-pressure wound therapy
  Arms: Negative-pressure wound therapy
Procedure: Conventional wound dressings — Conventional wound dressings
  Arms: Standard

SUMMARY:
There is a treatment method called negative-pressure wound therapy (NPWT) that is well established and used for the treatment of wounds. The method involves the application of a wound dressing through which a negative pressure is applied. Due to a plastic film overlaying the wound the risk of wound contamination is reduced. NPWT is considered to promote wound healing and prevent infection and has previously been used in the treatment of acute war associated wounds with satisfactory results. The aim of this study is to compare NPWT with conventional wound dressings in the treatment of war-associated extremity wounds and evaluate which method is more effective.

DETAILED DESCRIPTION:
Trial locations:

Médecins Sans Frontières/Doctors Without Borders (MSF) is one of the worlds leading independent organizations for medical humanitarian aid. MSF conducts an emergency trauma project in the Ministry of Health hospital in Ar Ramtha, Jordan, less than five kilometers from the border with Daraa governorate in Syria. A majority of patients within the project receive treatment for blast- and gunshot-related trauma wounds originating from the Syrian armed conflict. Within the project wound management has been difficult, often complicated by infection and antibiotic resistance. A need for wound therapy alternatives better than the conventional wound dressing method currently used has been identified.

Emergency hospital in Erbil, Iraq is a trauma hospital. Patients originate from armed conflicts in Mosul and the Iraqi Kurdistan region.

Background:

Extremity wounds and fractures constitute the majority of war-associated traumatic injuries, both for civilians (Aboutanos & Baker 1997) and combatants (Owens et al. 2007). Conflict-related injuries often result in soft and boney tissue being contaminated with foreign material, generally leading to secondary infection (Fares et al. 2013; Covey et al. 2000). Negative-pressure wound therapy (NPWT) is widely used in the treatment of wounds and is considered to promote wound healing and prevent infectious complications. The technique involves the application of a wound dressing through which a negative pressure is applied. Any wound and tissue fluid is drawn away from the area and collected into a canister. The risk of wound contamination is reduced by a plastic film overlaying the wound. NPWT is supported for use in a range of surgical applications, including after or in between debridements as a bridge to definite closure of soft tissue wounds (Krug et al. 2011). The technique has previously been used in the treatment of acute conflict-related wounds with satisfactory results (Machen 2006; Peck et al. 2007; Leininger et al. 2006).

Cochrane reviews of NPWT for the treatment of chronic wounds (Ubbink et al. 2008) and surgical wounds (Webster & Scuffham 2014) were inconclusive due to the lack of suitably powered, high-quality trials. A recent systematic review of randomized, controlled trials (RCTs) of NPWT for the treatment of acute and chronic wounds concluded there is a lack of evidence and that good RCTs are needed (Peinemann & Sauerland 2011). For the use in limb trauma, NPWT is considered suitable for complex soft tissue injuries (Bovill et al. 2008). NPWT appears to be an effective and safe adjunctive treatment of high-energy combat wounds but existing results are retrospective and lack follow-up (Hinck et al. 2010). The support of RCTs is needed to establish best treatment strategies.

Summary of potential risks and benefits:

Both treatment methods (NPWT and conventional dressings) are well established and used in Jordan for the treatment of acute and chronic wounds. As neither of the two treatment modalities are known to be better in terms of outcome neither patient group may be regarded as receiving preferential treatment. NPWT is generally considered a safe treatment method. Potential benefits are shortened healing time and fewer infectious complications. Potential risks are pain, mainly associated with dressing changes (Krasner 2002) and bleeding, predominantly minor bleeding from granulation tissue (Argenta, Louis Morykwas 1997). Conventional wound dressing has the potential benefit of being a safe treatment method used for many years. Since this method permits air into the wound there is a potential risk of contamination and the development of wound infection.

Objectives:

We aim to evaluate the efficacy and safety of NPWT in the treatment of traumatic extremity wounds in a context associated with a high level of contamination and infection.

Design:

A prospective, randomized, controlled trial comparing NPWT to conventional dressing methods in the treatment of conflict-related extremity wounds. Patients will continuously be included as they present at the emergency department of the hospital in Ar Ramtha.

Information for patients and consent:

Written and oral information in English and Arabic will be given to eligible participants. English versions of the participation information sheet and the consent form are provided as appendices to this document. Participants will be informed regarding their right to withdraw from the study and issues concerning confidentiality and the information sheet will remain with the participant. No incentives or inducements will be provided to any participant.

Eligible concomitant therapies:

Any signs of infection will be treated according to local standard protocols. Wounds in need of debridement will be debrided according to International Committee of the Red Cross (ICRC) war surgery protocols.

Interventions:

Patients randomly assigned to NPWT will receive treatment according to manufacturer treatment guidelines. Patients in the control group will be treated with conventional wound therapy according to local treatment protocols. In both groups dressing changes will be performed according to ICRC war surgery protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with extremity blast- or gunshot-wound(s). In case of multiple wounds the extremity wound with the estimated largest area is selected.

Exclusion Criteria:

* Wounds presenting >72 hours following initial trauma.
* Wounds that are considered ready for primary closure by suture or split-thickness skin graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Early wound closure | Day five +-1
  Wound closure, either by suture or split-thickness skin graft
Cost-effectiveness comparing outcomes from NPWT and standard treatment | Days (between 1 and 50)
  Costs from the health care provider's perspective will be used. Cost-effectiveness will be expressed in US dollars.

SECONDARY OUTCOMES:
Rate of wound healing | Days (between 1 and 50)
  Days to wound closure by suture or split-thickness skin graft
Wound infection | Days (between 1 and 50)
  Verified by either positive culture or clinical sign of infection, defined as purulent discharge
Time until wound is deemed no longer requiring professional care | Days (between 1 and 50)
Time to discharge | Days (between 1 and 50)
  Number of days to discharge
Quality of life aspects | Days five and eight
  Quality of life aspects including noise generated by the NPWT pump, movement impairment, skin irritation, odour, sleep quality, discomfort during dressing changes and pain
Full wound healing at follow-up | Day 30 following wound closure
  Full epithelialization
Septicaemia | Days (between 1 and 50)
  Septicaemia verified by positive blood culture
Mortality | Days (between 1 and 50)
  Death
Wound size ratio day fourteen | Day 14
  Wound size day fourteen divided by size day zero, i.e. wound healing rate after fourteen days
Number of surgeries | Days (between 1 and 50)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Malmstedt, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Emergency Hospital, Erbil, Kurdistan Region, Iraq
- Ar Ramtha Hospital, Ar Ramtha, Jordan

REFERENCES:
- [Result] Aboutanos MB, Baker SP. Wartime civilian injuries: epidemiology and intervention strategies. J Trauma. 1997 Oct;43(4):719-26. doi: 10.1097/00005373-199710000-00031. PMID 9356079
- [Result] Owens BD, Kragh JF Jr, Macaitis J, Svoboda SJ, Wenke JC. Characterization of extremity wounds in Operation Iraqi Freedom and Operation Enduring Freedom. J Orthop Trauma. 2007 Apr;21(4):254-7. doi: 10.1097/BOT.0b013e31802f78fb. PMID 17414553
- [Result] Fares Y, El-Zaatari M, Fares J, Bedrosian N, Yared N. Trauma-related infections due to cluster munitions. J Infect Public Health. 2013 Dec;6(6):482-6. doi: 10.1016/j.jiph.2013.05.006. Epub 2013 Jul 31. PMID 23999350
- [Result] Covey DC, Lurate RB, Hatton CT. Field hospital treatment of blast wounds of the musculoskeletal system during the Yugoslav civil war. J Orthop Trauma. 2000 May;14(4):278-86; discussion 277. doi: 10.1097/00005131-200005000-00010. PMID 10898201
- [Result] Krug E, Berg L, Lee C, Hudson D, Birke-Sorensen H, Depoorter M, Dunn R, Jeffery S, Duteille F, Bruhin A, Caravaggi C, Chariker M, Dowsett C, Ferreira F, Martinez JM, Grudzien G, Ichioka S, Ingemansson R, Malmsjo M, Rome P, Vig S, Runkel N, Martin R, Smith J; International Expert Panel on Negative Pressure Wound Therapy [NPWT-EP]. Evidence-based recommendations for the use of Negative Pressure Wound Therapy in traumatic wounds and reconstructive surgery: steps towards an international consensus. Injury. 2011 Feb;42 Suppl 1:S1-12. doi: 10.1016/S0020-1383(11)00041-6. PMID 21316515
- [Result] Machen S. Management of traumatic war wounds using vacuum-assisted closure dressings in an austere environment. US Army Med Dep J. 2007 Jan-Mar:17-23. PMID 20084702
- [Result] Peck MA, Clouse WD, Cox MW, Bowser AN, Eliason JL, Jenkins DH, Smith DL, Rasmussen TE. The complete management of extremity vascular injury in a local population: a wartime report from the 332nd Expeditionary Medical Group/Air Force Theater Hospital, Balad Air Base, Iraq. J Vasc Surg. 2007 Jun;45(6):1197-204; discussion 1204-5. doi: 10.1016/j.jvs.2007.02.003. PMID 17543685
- [Result] Leininger BE, Rasmussen TE, Smith DL, Jenkins DH, Coppola C. Experience with wound VAC and delayed primary closure of contaminated soft tissue injuries in Iraq. J Trauma. 2006 Nov;61(5):1207-11. doi: 10.1097/01.ta.0000241150.15342.da. PMID 17099530
- [Result] Ubbink DT, Westerbos SJ, Evans D, Land L, Vermeulen H. Topical negative pressure for treating chronic wounds. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD001898. doi: 10.1002/14651858.CD001898.pub2. PMID 18646080
- [Result] Webster J, Scuffham P, Stankiewicz M, Chaboyer WP. Negative pressure wound therapy for skin grafts and surgical wounds healing by primary intention. Cochrane Database Syst Rev. 2014 Oct 7;(10):CD009261. doi: 10.1002/14651858.CD009261.pub3. PMID 25287701
- [Result] Peinemann F, Sauerland S. Negative-pressure wound therapy: systematic review of randomized controlled trials. Dtsch Arztebl Int. 2011 Jun;108(22):381-9. doi: 10.3238/arztebl.2011.0381. Epub 2011 Jun 3. PMID 21712971
- [Result] Bovill E, Banwell PE, Teot L, Eriksson E, Song C, Mahoney J, Gustafsson R, Horch R, Deva A, Whitworth I; International Advisory Panel on Topical Negative Pressure. Topical negative pressure wound therapy: a review of its role and guidelines for its use in the management of acute wounds. Int Wound J. 2008 Oct;5(4):511-29. doi: 10.1111/j.1742-481X.2008.00437.x. Epub 2008 Sep 19. PMID 18808432
- [Result] Hinck D, Franke A, Gatzka F. Use of vacuum-assisted closure negative pressure wound therapy in combat-related injuries--literature review. Mil Med. 2010 Mar;175(3):173-81. doi: 10.7205/milmed-d-09-00075. PMID 20358706
- [Result] Krasner DL. Managing wound pain in patients with vacuum-assisted closure devices. Ostomy Wound Manage. 2002 May;48(5):38-43. PMID 12046489
- [Result] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Derived] Haque G, Haweizy R, Bashaireh K, Malmstedt J, Alga A. Impact of injury mechanism on early wound closure in patients with acute conflict-related extremity wounds: A prospective cohort analysis from two civilian hospitals in Iraq and Jordan. World J Surg. 2024 Aug;48(8):1822-1828. doi: 10.1002/wjs.12276. Epub 2024 Jul 5. PMID 38970237
- [Derived] Alga A, Lofgren J, Haweizy R, Bashaireh K, Wong S, Forsberg BC, von Schreeb J, Malmstedt J. Cost analysis of negative-pressure wound therapy versus standard treatment of acute conflict-related extremity wounds within a randomized controlled trial. World J Emerg Surg. 2022 Feb 10;17(1):9. doi: 10.1186/s13017-022-00415-1. PMID 35144650
- [Derived] Alga A, Haweizy R, Bashaireh K, Wong S, Lundgren KC, von Schreeb J, Malmstedt J. Negative pressure wound therapy versus standard treatment in patients with acute conflict-related extremity wounds: a pragmatic, multisite, randomised controlled trial. Lancet Glob Health. 2020 Mar;8(3):e423-e429. doi: 10.1016/S2214-109X(19)30547-9. PMID 32087175
- [Derived] Alga A, Wong S, Haweizy R, Conneryd Lundgren K, von Schreeb J, Malmstedt J. Negative-Pressure Wound Therapy Versus Standard Treatment of Adult Patients With Conflict-Related Extremity Wounds: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Nov 26;7(11):e12334. doi: 10.2196/12334. PMID 30478024